CLINICAL TRIAL: NCT04513080
Title: Message-Based Psychotherapy and Digital Treatment Sequences for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Talkspace (Industry)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Aarthi Padmanabhan, Senior Director of Research, Talkspace
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00010391
Record Dates: First submitted 2020-08-09; First posted 2020-08-14 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Study Adherence; Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Intervention Model Description: Phase 1 will test the effectiveness of two forms of participant retention methods into a SMART (sequential, multiple assignment, randomized). In Phase 1, participants (n=200) will be randomized to an incentive level and then randomized to treatment arms. Phase 2 (n=1000) will be the subsequent SMART design comparing message-based psychotherapy (MBP) to video-chat psychotherapy (VCP) in level 1 and for those who do not respond to care after 6 weeks, those participants will be randomized to either MBP+monthly VCP or MBP+weekly VCP.
  Arms/Interventions have been adjusted to align with the results for the Phase 2 SMART.
Who Masked: Outcomes Assessor
Masking Description: In Phase 1, participants will be masked to the incentive condition to which they are randomized but will be aware of which treatment condition they are receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- Phase 2: Message-Based Psychotherapy (MBP; Level 1 and Level 2) (Experimental): Phase 2 participants who respond to Message-Based Psychotherapy (MBP; Level 1) by 5 weeks of care will continue in this condition from weeks 6 to 12 (MBP; Level 2).
  Interventions: Behavioral: Message-Based Psychotherapy (MBP)
- Phase 2: Video-Chat Psychotherapy (VCP; Level 1 and Level 2) (Experimental): Phase 2 participants who respond to Video-Chat Psychotherapy (VCP; Level 1) by 5 weeks of care will continue in this condition from weeks 6 to 12 (VCP; Level 2). VCP consists of weekly psychotherapy appointments that last between 30-45 minutes.
  Interventions: Behavioral: Video-Chat Psychotherapy (VCP)
- Phase 2: MBP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2) (Experimental): Phase 2: This arm includes participants in MBP (Level 1) who do not respond to treatment by week 5. The Premium Plan intervention consists of MBP with monthly VCP (Level 2). The Premium Plan allows patients unlimited MBP and once a month, 30-45 minute video chat with the same therapist. This intervention will serve as one of two Level 2 conditions for participants who do not respond to MBP or VCP alone by week 5.
  Interventions: Behavioral: Message-Based Psychotherapy (MBP); Behavioral: Message-Based Psychotherapy with Monthly Video-Chat Psychotherapy
- Phase 2: MBP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2) (Experimental): Phase 2: This arm includes participants in MBP (Level 1) who do not respond to treatment by week 5. The Ultimate Plan intervention consists of MBP with weekly VCP (Level 2). The Ultimate Plan allows patients unlimited MBP and weekly, 30-45 minute video chat with the same therapist. This intervention will serve as one of two Level 2 conditions for participants who do not respond to MBP or VCP alone by week 5.
  Interventions: Behavioral: Message-Based Psychotherapy (MBP); Behavioral: Message-Based Psychotherapy with Weekly Video-Chat Psychotherapy
- Phase 2: VCP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2) (Experimental): Phase 2: This arm includes participants in VCP (Level 1) who do not respond to treatment by week 5. The Premium Plan intervention consists of MBP with monthly VCP (Level 2). The Premium Plan allows patients unlimited MBP and once a month, 30-45 minute video chat with the same therapist. This intervention will serve as one of two Level 2 conditions for participants who do not respond to MBP or VCP alone by week 5.
  Interventions: Behavioral: Video-Chat Psychotherapy (VCP); Behavioral: Message-Based Psychotherapy with Monthly Video-Chat Psychotherapy
- Phase 2: VCP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2) (Experimental): Phase 2: This arm includes participants in VCP (Level 1) who do not respond to treatment by week 5. The Ultimate Plan intervention consists of MBP with weekly VCP (Level 2). The Ultimate Plan allows patients unlimited MBP and weekly, 30-45 minute video chat with the same therapist. This intervention will serve as one of two Level 2 conditions for participants who do not respond to MBP or VCP alone by week 5.
  Interventions: Behavioral: Video-Chat Psychotherapy (VCP); Behavioral: Message-Based Psychotherapy with Weekly Video-Chat Psychotherapy
- Phase 1: High Monetary Incentive (HMI) + VCP (Level 1 and Level 2) (Experimental): Phase 1 participants who respond to VCP (Level 1) by 5 weeks of care will continue in this condition from weeks 6 to 12 (VCP; Level 2). Participants in the High Monetary Incentive (HMI) arm received a total of $125 for completing 12 weeks of assessments.
  Interventions: Behavioral: Video-Chat Psychotherapy (VCP); Behavioral: High Monetary Incentive (HMI)
- Phase 1: High Monetary Incentive (HMI) + MBP (Level 1 and Level 2) (Experimental): Phase 1 participants who respond to MBP (Level 1) by 5 weeks of care will continue in this condition from weeks 6 to 12 (MBP; Level 2). Participants in the High Monetary Incentive (HMI) arm received a total of $125 for completing 12 weeks of assessments.
  Interventions: Behavioral: Message-Based Psychotherapy (MBP); Behavioral: High Monetary Incentive (HMI)
- Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1 and Level 2) (Experimental): Phase 1 participants who respond to VCP (Level 1) by 5 weeks of care will continue in this condition from weeks 6 to 12 (VCP; Level 2). Participants in the Low Monetary and Alternative Incentive (LMAI) arm received a total of $75 for completing 12 weeks of assessments, messages of encouragement for completing daily assessments, and weekly texts showing participants their clinical improvement and assessment completion rate.
  Interventions: Behavioral: Video-Chat Psychotherapy (VCP); Behavioral: Low Monetary and Alternative Incentive (LMAI)
- Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1 and Level 2) (Experimental): Phase 1 participants who respond to MBP (Level 1) by 5 weeks of care will continue in this condition from weeks 6 to 12 (MBP; Level 2). Participants in the Low Monetary and Alternative Incentive (LMAI) arm received a total of $75 for completing 12 weeks of assessments, messages of encouragement for completing daily assessments, and weekly texts showing participants their clinical improvement and assessment completion rate.
  Interventions: Behavioral: Message-Based Psychotherapy (MBP); Behavioral: Low Monetary and Alternative Incentive (LMAI)
- Phase 1: HMI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) (Experimental): Phase 1: This arm includes participants in HMI + VCP (Level 1) who do not respond to treatment by week 5. The Augmentation Arm consists of MBP with weekly VCP (Level 2). Participants will have access to unlimited MBP and will be able to schedule weekly, 30-45 minute video chat with the same therapist. This intervention will serve as one of two conditions for participants who do not respond to MBP or VCP alone by week 5.
  Interventions: Behavioral: Message-Based Psychotherapy with Weekly Video-Chat Psychotherapy; Behavioral: High Monetary Incentive (HMI)
- Phase 1: HMI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2) (Experimental): Phase 1: This arm includes participants in HMI + VCP (Level 1) who do not respond to treatment by week 5. The Switch Arm consists of MBP with monthly VCP (Level 2). Patients have access to unlimited MBP and once a month, 30-45 minute video chat with the same therapist. This intervention will serve as one of two conditions for participants who do not respond to MBP or VCP alone by week 5.
  Interventions: Behavioral: Message-Based Psychotherapy with Monthly Video-Chat Psychotherapy; Behavioral: High Monetary Incentive (HMI)
- Phase 1: HMI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) (Experimental): Phase 1: This arm includes participants in HMI + MBP (Level 1) who do not respond to treatment by week 5. The Augmentation Arm consists of MBP with weekly VCP (Level 2). Participants will have access to unlimited MBP and will be able to schedule weekly, 30-45 minute video chat with the same therapist. This intervention will serve as one of two conditions for participants who do not respond to MBP or VCP alone by week 5.
  Interventions: Behavioral: Message-Based Psychotherapy with Weekly Video-Chat Psychotherapy; Behavioral: High Monetary Incentive (HMI)
- Phase 1: HMI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2) (Experimental): Phase 1: This arm includes participants in HMI + MBP (Level 1) who do not respond to treatment by week 5. The Minimal Augmentation arm consists of MBP with monthly VCP (Level 2). Patients have access to unlimited MBP and once a month, 30-45 minute video chat with the same therapist. This intervention will serve as one of two conditions for participants who do not respond to MBP or VCP alone by week 5.
  Interventions: Behavioral: Message-Based Psychotherapy with Monthly Video-Chat Psychotherapy; Behavioral: High Monetary Incentive (HMI)
- Phase 1: LMAI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) (Experimental): Phase 1: This arm includes participants in LMAI + VCP (Level 1) who do not respond to treatment by week 5. The Augmentation Arm consists of MBP with weekly VCP (Level 2). Participants will have access to unlimited MBP and will be able to schedule weekly, 30-45 minute video chat with the same therapist. This intervention will serve as one of two conditions for participants who do not respond to MBP or VCP alone by week 5.
  Interventions: Behavioral: Message-Based Psychotherapy with Weekly Video-Chat Psychotherapy; Behavioral: Low Monetary and Alternative Incentive (LMAI)
- Phase 1: LMAI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2) (Experimental): Phase 1: This arm includes participants in LMAI + VCP (Level 1) who do not respond to treatment by week 5. The Switch Arm consists of MBP with monthly VCP (Level 2). Patients have access to unlimited MBP and once a month, 30-45 minute video chat with the same therapist. This intervention will serve as one of two conditions for participants who do not respond to MBP or VCP alone by week 5.
  Interventions: Behavioral: Message-Based Psychotherapy with Monthly Video-Chat Psychotherapy; Behavioral: Low Monetary and Alternative Incentive (LMAI)
- Phase 1: LMAI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) (Experimental): Phase 1: This arm includes participants in LMAI + MBP (Level 1) who do not respond to treatment by week 5. The Augmentation Arm consists of MBP with weekly VCP (Level 2). Participants will have access to unlimited MBP and will be able to schedule weekly, 30-45 minute video chat with the same therapist. This intervention will serve as one of two conditions for participants who do not respond to MBP or VCP alone by week 5.
  Interventions: Behavioral: Message-Based Psychotherapy with Weekly Video-Chat Psychotherapy; Behavioral: Low Monetary and Alternative Incentive (LMAI)
- Phase 1: LMAI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2) (Experimental): Phase 1: This arm includes participants in LMAI + MBP (Level 1) who do not respond to treatment by week 5. The Minimal Augmentation arm consists of MBP with monthly VCP (Level 2). Patients have access to unlimited MBP and once a month, 30-45 minute video chat with the same therapist. This intervention will serve as one of two conditions for participants who do not respond to MBP or VCP alone by week 5.
  Interventions: Behavioral: Message-Based Psychotherapy with Monthly Video-Chat Psychotherapy; Behavioral: Low Monetary and Alternative Incentive (LMAI)

INTERVENTIONS:
Behavioral: Video-Chat Psychotherapy (VCP) — Video-Chat Psychotherapy (VCP) consists of weekly psychotherapy appointments that last between 30-45 minutes. These sessions are conducted using Agora, a secure, HIPAA-compliant video conferencing service that is seamlessly integrated into the Talkspace platform application. Therapists will provide evidence-based treatments for depression and anxiety.
  Arms: Phase 1: High Monetary Incentive (HMI) + VCP (Level 1 and Level 2); Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1 and Level 2); Phase 2: VCP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2); Phase 2: VCP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2); Phase 2: Video-Chat Psychotherapy (VCP; Level 1 and Level 2)
Behavioral: Message-Based Psychotherapy (MBP) — Message-Based Psychotherapy (MBP) allows patients to chat with an assigned licensed therapist as frequently as they wish. After consumers complete an intake and select a therapist, the consumer can begin chatting with their therapist right away, and as often as they wish. Therapists respond to text within 15 minutes to an hour during office hours, and within 14 hours outside of office hours. Thus, MBP is not fully synchronous. This enables therapists to deliver care to a larger number of patients than is possible under synchronous methods by disentangling the therapist's time from the patient's time to respond. It also has the potential to improve quality as it gives the therapist time to think through the most effective response and intervention. MBP will be based on CBT, PST or IPT intervention strategies.
  Arms: Phase 1: High Monetary Incentive (HMI) + MBP (Level 1 and Level 2); Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1 and Level 2); Phase 2: MBP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2); Phase 2: MBP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2); Phase 2: Message-Based Psychotherapy (MBP; Level 1 and Level 2)
Behavioral: Message-Based Psychotherapy with Monthly Video-Chat Psychotherapy — Message-Based Psychotherapy (MBP) with monthly Video-Chat Psychotherapy (VCP) allows patients unlimited texting with their therapist and once a month, 30-45 minute video chat with the same therapist. Therapist and participants schedule their video chat appointment to occur at once a month interval during therapist office hours. The content of these sessions, as well as the MBP portion of care, will be based on CBT, PST or IPT. In Phase 1, this is referred to as "Switch Arm" (for participants assigned to VCP at baseline) or "Minimal Augmentation" (for participants assigned to MBP at baseline). In Phase 2, this is referred to as the "Premium Plan".
  Arms: Phase 1: HMI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2); Phase 1: HMI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2); Phase 1: LMAI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2); Phase 1: LMAI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2); Phase 2: MBP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2); Phase 2: VCP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2)
Behavioral: Message-Based Psychotherapy with Weekly Video-Chat Psychotherapy — Message-Based Psychotherapy (MBP) with weekly Video-Chat Psychotherapy (VCP) allows patients access to both unlimited MBP, but will be able to schedule weekly, 30-45 minute video chat with the same therapist. Therapists will provide care based on CBT, PST or IPT. In Phase 1, this is referred to as the "Augmentation Arm". In Phase 2, this is referred to as the "Ultimate Plan."
  Arms: Phase 1: HMI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2); Phase 1: HMI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2); Phase 1: LMAI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2); Phase 1: LMAI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2); Phase 2: MBP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2); Phase 2: VCP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2)
Behavioral: High Monetary Incentive (HMI) — Participants in the traditional, high monetary incentive arm will receive a total of $125 for completing 12 weeks of assessments.
  Arms: Phase 1: HMI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2); Phase 1: HMI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2); Phase 1: HMI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2); Phase 1: HMI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2); Phase 1: High Monetary Incentive (HMI) + MBP (Level 1 and Level 2); Phase 1: High Monetary Incentive (HMI) + VCP (Level 1 and Level 2)
Behavioral: Low Monetary and Alternative Incentive (LMAI) — Participants in the Low Monetary and Alternative Incentive (LMAI) arm received a total of $75 for completing 12 weeks of assessments, messages of encouragement for completing daily assessments, and weekly texts showing participants their clinical improvement and assessment completion rate.
  Arms: Phase 1: LMAI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2); Phase 1: LMAI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2); Phase 1: LMAI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2); Phase 1: LMAI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2); Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1 and Level 2); Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1 and Level 2)

SUMMARY:
This partnership between Talkspace and the University of Washington (UW) ALACRITY Center will determine how effective unlimited text-based psychotherapy for depression is when compared to once-a-week psychotherapy. This study will also determine what the best treatment options are for people who are not responding well to either unlimited texting or weekly psychotherapy. The results of this study will be a new product version of message-based care that can tailor psychotherapy intensity based on the needs of future consumers with depression.

DETAILED DESCRIPTION:
This is a fast track Small Business Innovation Research (SBIR) proposal that will (1) test the effectiveness of daily, message-based psychotherapy (MBP) for depression, compared to traditionally delivered, video-chat psychotherapy (VCP) and (2) develop an evidence-based treatment sequence for those who do not respond to either daily MBP or VCP.

Phase 1 consists of a pilot study to determine the best incentive model to retain a sample of people 18 years old and older with depression into a SMART trial. Information from this pilot will inform the retention strategy for Phase 2.

Phase 2 is a 12-week, randomized clinical trial using a SMART design to test the following aims: 1. Determine the relative effectiveness of daily MBP compared to weekly VCP in treating symptoms of depression and improving social functioning; 2. For those who fail to respond to 6 weeks of weekly VCP only, determine whether the addition of daily messaging, or a switch to monthly video-chat plus daily messaging improves depression and functional outcomes; and 3. For those who fail to respond to 6 weeks of daily MBP, whether the addition of monthly video-chat or weekly video-chat improves outcomes. Participants will provide data on mood, activity, and functioning, and we will collect data on use of treatment (texts and sessions), and working alliance.

ELIGIBILITY:
Inclusion and exclusion criteria are the same for Phase 1 and Phase 2.

Inclusion Criteria:

* 18 years old or older
* English or Spanish speaking
* Live in the United States
* Score of 10 or greater on the Patient Health Questionnaire-9 (PHQ-9) screening
* Receive a diagnosis of depression from a Talkspace intake clinician

Exclusion Criteria:

* Under the age of 18
* Non-English or Spanish speaking
* Do not meet criteria for a depressive disorder
* Participants with active suicidal ideation or with a primary diagnosis of psychosis will also be excluded and referred to intensive care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1184 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2024-01-14 (Actual); Study Completion 2024-01-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Talkspace, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Quantitative data is available upon reasonable request with a fully executed Data Use Agreement with Talkspace.

REFERENCES:
- [Derived] Pullmann MD, Rouvere J, Raue PJ, Griffith Fillipo IR, Mosser BA, Heagerty PJ, Fridling-Cook N, Padmanabhan A, Hull TD, Arean PA. Message-Based vs Video-Based Psychotherapy for Depression: A Randomized Clinical Trial. JAMA Netw Open. 2025 Oct 1;8(10):e2540065. doi: 10.1001/jamanetworkopen.2025.40065. PMID 41165707
- [Derived] Arean P, Hull D, Pullmann MD, Heagerty PJ. Protocol for a sequential, multiple assignment, randomised trial to test the effectiveness of message-based psychotherapy for depression compared with telepsychotherapy. BMJ Open. 2021 Nov 2;11(11):e046958. doi: 10.1136/bmjopen-2020-046958. PMID 34728440

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Baseline to Week 5: "Participated in the Intervention" includes the analytic sample for Level 1 analyses. "Completed" is defined as participants evaluated for Level 2 randomization.
  Week 6 to Week 12: Phase 1 "Completed" is defined as having completed the PHQ-9 at any time between weeks 6 to 12. Phase 2 "Completed" is defined as having completed outcome measures between weeks 6 to 12.
Pre-assignment Details: The Participant Flow below shows arms by combination of Level 1 and Level 2 conditions. Sample sizes from baseline to week 5 apply to Level 1 conditions. Sample sizes from week 6 to week 12 apply to Level 2 conditions. Therefore, sample sizes for arms including Level 2 conditions from baseline to week 5 are 0.
Groups:
- Phase 2: MBP (Level 1) to Preimum Plan (MBP with monthly VCP; Level 2): Phase 2: This arm includes participants in MBP (Level 1) who do not respond to treatment by week 5. The Premium Plan intervention consists of MBP with monthly VCP (Level 2). The Premium Plan allows patients unlimited MBP and once a month, 30-45 minute video chat with the same therapist. This intervention will serve as one of two Level 2 conditions for participants who do not respond to MBP or VCP alone by week 5.
- Phase 2: VCP (Level 1) to Preimum Plan (MBP with monthly VCP; Level 2): Phase 2: This arm includes participants in VCP (Level 1) who do not respond to treatment by week 5. The Premium Plan intervention consists of MBP with monthly VCP (Level 2). The Premium Plan allows patients unlimited MBP and once a month, 30-45 minute video chat with the same therapist. This intervention will serve as one of two Level 2 conditions for participants who do not respond to MBP or VCP alone by week 5.
Period: Baseline to Week 5 - Level 1
Arm/Group | Phase 2: Message-Based Psychotherapy (MBP; Level 1 and Level 2) | Phase 2: Video-Chat Psychotherapy (VCP; Level 1 and Level 2) | Phase 2: MBP (Level 1) to Preimum Plan (MBP with monthly VCP; Level 2) | Phase 2: MBP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2) | Phase 2: VCP (Level 1) to Preimum Plan (MBP with monthly VCP; Level 2) | Phase 2: VCP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2) | Phase 1: High Monetary Incentive (HMI) + VCP (Level 1 and Level 2) | Phase 1: High Monetary Incentive (HMI) + MBP (Level 1 and Level 2) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1 and Level 2) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1 and Level 2) | Phase 1: HMI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: HMI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2) | Phase 1: HMI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: HMI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2) | Phase 1: LMAI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: LMAI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2) | Phase 1: LMAI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: LMAI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2)
Started | 485 | 484 | 0 | 0 | 0 | 0 | 55 | 54 | 52 | 54 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Participated in the Intervention | 423 | 427 | 0 | 0 | 0 | 0 | 55 | 54 | 52 | 54 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Evaluated for Level 2 randomization) | 363 | 336 | 0 | 0 | 0 | 0 | 37 | 37 | 37 | 46 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 122 | 148 | 0 | 0 | 0 | 0 | 18 | 17 | 15 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Week 6 to Week 12 - Level 2
Arm/Group | Phase 2: Message-Based Psychotherapy (MBP; Level 1 and Level 2) | Phase 2: Video-Chat Psychotherapy (VCP; Level 1 and Level 2) | Phase 2: MBP (Level 1) to Preimum Plan (MBP with monthly VCP; Level 2) | Phase 2: MBP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2) | Phase 2: VCP (Level 1) to Preimum Plan (MBP with monthly VCP; Level 2) | Phase 2: VCP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2) | Phase 1: High Monetary Incentive (HMI) + VCP (Level 1 and Level 2) | Phase 1: High Monetary Incentive (HMI) + MBP (Level 1 and Level 2) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1 and Level 2) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1 and Level 2) | Phase 1: HMI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: HMI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2) | Phase 1: HMI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: HMI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2) | Phase 1: LMAI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: LMAI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2) | Phase 1: LMAI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: LMAI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2)
Started | 105 | 93 | 114 | 144 | 126 | 117 | 15 | 11 | 12 | 17 | 10 | 12 | 13 | 13 | 12 | 13 | 13 | 16
Completed | 99 | 88 | 108 | 133 | 115 | 107 | 12 | 11 | 9 | 15 | 9 | 9 | 12 | 13 | 9 | 12 | 12 | 11
Not Completed | 6 | 5 | 6 | 11 | 11 | 10 | 3 | 0 | 3 | 2 | 1 | 3 | 1 | 0 | 3 | 1 | 1 | 5

BASELINE CHARACTERISTICS:
Population: All participants randomized to a Level 1 condition who participated in the intervention.
Groups:
- Phase 2: Message-Based Psychotherapy (MBP; Level 1): Message-Based Psychotherapy (MBP) allows patients to chat with an assigned licensed therapist as frequently as they wish. After consumers complete an intake and select a therapist, the consumer can begin chatting with their therapist right away, and as often as they wish. Therapists respond to text within 15 minutes to an hour during office hours, and within 14 hours outside of office hours. Thus, MBP is not fully synchronous. This enables therapists to deliver care to a larger number of patients than is possible under synchronous methods by disentangling the therapist's time from the patient's time to respond. It also has the potential to improve quality as it gives the therapist time to think through the most effective response and intervention. MBP will be based on CBT, PST or IPT intervention strategies.
- Phase 2: Video-Chat Psychotherapy (VCP; Level 1): Video-Chat Psychotherapy (VCP) consists of weekly psychotherapy appointments that last between 30-45 minutes. These sessions are conducted using Agora, a secure, HIPAA-compliant video conferencing service that is seamlessly integrated into the Talkspace platform application. Therapists will provide evidence-based treatments for depression and anxiety.
- Phase 1: High Monetary Incentive (HMI) + VCP (Level 1): Participants in the High Monetary Incentive (HMI) arm received a total of $125 for completing 12 weeks of assessments. Video-Chat Psychotherapy (VCP) consists of weekly psychotherapy appointments that last between 30-45 minutes. These sessions are conducted using Agora, a secure, HIPAA-compliant video conferencing service that is seamlessly integrated into the Talkspace platform application. Therapists will provide evidence-based treatments for depression and anxiety.
- Phase 1: High Monetary Incentive (HMI) + MBP (Level 1): Participants in the High Monetary Incentive (HMI) arm received a total of $125 for completing 12 weeks of assessments. Message-Based Psychotherapy (MBP) allows patients to chat with an assigned licensed therapist as frequently as they wish. After consumers complete an intake and select a therapist, the consumer can begin chatting with their therapist right away, and as often as they wish. Therapists respond to text within 15 minutes to an hour during office hours, and within 14 hours outside of office hours. Thus, MBP is not fully synchronous. This enables therapists to deliver care to a larger number of patients than is possible under synchronous methods by disentangling the therapist's time from the patient's time to respond. It also has the potential to improve quality as it gives the therapist time to think through the most effective response and intervention. MBP will be based on CBT, PST or IPT intervention strategies.
- Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1): Participants in the Low Monetary and Alternative Incentive (LMAI) arm received a total of $75 for completing 12 weeks of assessments, messages of encouragement for completing daily assessments, and weekly texts showing participants their clinical improvement and assessment completion rate. Video-Chat Psychotherapy (VCP) consists of weekly psychotherapy appointments that last between 30-45 minutes. These sessions are conducted using Agora, a secure, HIPAA-compliant video conferencing service that is seamlessly integrated into the Talkspace platform application. Therapists will provide evidence-based treatments for depression and anxiety.
- Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1): Participants in the Low Monetary and Alternative Incentive (LMAI) arm received a total of $75 for completing 12 weeks of assessments, messages of encouragement for completing daily assessments, and weekly texts showing participants their clinical improvement and assessment completion rate. Message-Based Psychotherapy (MBP) allows patients to chat with an assigned licensed therapist as frequently as they wish. After consumers complete an intake and select a therapist, the consumer can begin chatting with their therapist right away, and as often as they wish. Therapists respond to text within 15 minutes to an hour during office hours, and within 14 hours outside of office hours. Thus, MBP is not fully synchronous. This enables therapists to deliver care to a larger number of patients than is possible under synchronous methods by disentangling the therapist's time from the patient's time to respond. It also has the potential to improve quality as it gives the therapist time to think through the most effective response and intervention. MBP will be based on CBT, PST or IPT intervention strategies.
- Total: Total of all reporting groups
Arm/Group | Phase 2: Message-Based Psychotherapy (MBP; Level 1) | Phase 2: Video-Chat Psychotherapy (VCP; Level 1) | Phase 1: High Monetary Incentive (HMI) + VCP (Level 1) | Phase 1: High Monetary Incentive (HMI) + MBP (Level 1) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1) | Total
Number analyzed (Participants) | 423 | 427 | 55 | 54 | 52 | 54 | 1065
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Includes participants who participated in the intervention.
  years
    Phase 2: number analyzed (Participants) | 423 | 427 | 0 | 0 | 0 | 0 | 850
    Phase 2 | 33.4 (10.1) | 34.1 (10.9) |  |  |  |  | 33.8 (10.5)
    Phase 1: number analyzed (Participants) | 0 | 0 | 55 | 54 | 52 | 54 | 215
    Phase 1 |  |  | 31.25 (10.35) | 29.20 (10.04) | 29.48 (8.89) | 28.91 (8.86) | 29.72 (9.54)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 116 | 115 | 3 | 8 | 10 | 9 | 261
  Gender: Female | 275 | 287 | 47 | 44 | 38 | 42 | 733
  Gender: Other | 27 | 23 | 3 | 2 | 4 | 3 | 62
  Gender: Unknown or not reported | 5 | 2 | 2 | 0 | 0 | 0 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62 | 58 | 15 | 16 | 16 | 18 | 185
  Not Hispanic or Latino | 351 | 362 | 39 | 36 | 36 | 34 | 858
  Unknown or Not Reported | 10 | 7 | 1 | 2 | 0 | 2 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian/Alaskan Native | 1 | 5 | 0 | 0 | 0 | 0 | 6
  Race: Asian | 24 | 21 | 3 | 4 | 5 | 5 | 62
  Race: Black or African American | 97 | 93 | 3 | 3 | 7 | 7 | 210
  Race: Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Race: White or Caucasian | 259 | 253 | 33 | 34 | 31 | 30 | 640
  Race: Prefer to self describe | 9 | 9 | 5 | 3 | 3 | 4 | 33
  Race: Prefer not to say | 6 | 10 | 2 | 4 | 0 | 1 | 23
  Race: Multiple races | 22 | 33 | 9 | 6 | 6 | 7 | 83
  Race: Unknown or not reported | 5 | 2 | 0 | 0 | 0 | 0 | 7
Patient Health Questionnaire-9 (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire-9 (PHQ-9) consists of 9 depression items and one disability item. Each time is associated with a Diagnostic and Statistical Manual (DMS) symptom of depression, which the participant rates whether or not they have experienced the symptom over the last two weeks, with severity rating of 0-3. It is one of the few measures that is brief (it takes less than one minute to give) and has been found to have excellent sensitivity to change over time. Total scores range from 0-27, with higher scores indicating greater severity of depression. Population: Includes participants who provided data at baseline.
  units on a scale
    Phase 2: number analyzed (Participants) | 423 | 427 | 0 | 0 | 0 | 0 | 850
    Phase 2 | 14.98 (4.75) | 15.00 (4.84) |  |  |  |  | 14.99 (4.79)
    Phase 1: number analyzed (Participants) | 0 | 0 | 47 | 49 | 50 | 50 | 196
    Phase 1 |  |  | 17.45 (3.83) | 18.22 (4.47) | 16.76 (4.60) | 16.22 (4.55) | 17.15 (4.41)

OUTCOME MEASURES:

1. Primary Outcome: Change in Neuro-QOL - Ability to Participate in Social Roles and Activities
Description: Neuro-Quality of Life v1.0 (Neuro-QOL). The Neuro-QOL Ability to Participate in Social Roles and Activities short form item bank is an 8-item patient-rated measure of social functioning. Items focus on difficulty participating in social, family, and work activities, and are rated on a 1 to 5 scale for a total score between 8 and 40. Neuro-QOL scores were transformed into t-scores per the scoring manual; after transformation, total scores range from 24.1 to 60.2. Transformed scores are reported. Higher scores indicate less difficulty participating in social roles and activities. The Neuro-QOL was not distributed in Phase 1.
Time Frame: Change from Baseline Neuro-QOL at 6 weeks and 12 weeks after treatment starts
Population: Phase 2 participants contributing data at baseline, week 6, or week 12. Overall number of participants analyzed includes total number of participants who contributed data at any relevant timepoint.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Phase 2: Message-Based Psychotherapy (MBP; Level 1) | Phase 2: Video-Chat Psychotherapy (VCP; Level 1)
Number analyzed (Participants) | 393 | 402
T-score
  Baseline: number analyzed (Participants) | 388 | 401
  Baseline | 39.55 (3.93) | 39.57 (4.55)
  Week 6: number analyzed (Participants) | 338 | 300
  Week 6 | 41.65 (4.95) | 42.07 (5.47)
  Week 12: number analyzed (Participants) | 305 | 293
  Week 12 | 43.39 (6.50) | 43.11 (6.68)
Statistical Analysis 1: Comparison: Phase 2: Message-Based Psychotherapy (MBP; Level 1) vs Phase 2: Video-Chat Psychotherapy (VCP; Level 1); Mean difference comparing difference in average scores from baseline to week 6; Test type: Superiority; Mean Difference (Final Values) = 0.4
Statistical Analysis 2: Comparison: Phase 2: Message-Based Psychotherapy (MBP; Level 1) vs Phase 2: Video-Chat Psychotherapy (VCP; Level 1); Mean difference comparing difference in average scores from week 6 to week 12; Test type: Superiority; Mean Difference (Final Values) = 0.7

2. Primary Outcome: Change in Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire-9 (PHQ-9) consists of 9 depression items and one disability item. Each time is associated with a Diagnostic and Statistical Manual (DMS) symptom of depression, which the participant rates whether or not they have experienced the symptom over the last two weeks, with severity rating of 0-3. It is one of the few measures that is brief (it takes less than one minute to give) and has been found to have excellent sensitivity to change over time. Total scores range from 0-27, with higher scores indicating greater severity of depression.
Time Frame: Change from Baseline PHQ-9 at 6 weeks and 12 weeks after treatment starts
Population: All participants randomized to a Level 2 condition contributing data at baseline, week 6, or week 12. Overall number of participants analyzed includes total number of participants who contributed data at any relevant timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 2: Message-Based Psychotherapy (MBP; Level 1 and Level 2) | Phase 2: Video-Chat Psychotherapy (VCP; Level 1 and Level 2) | Phase 2: MBP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2) | Phase 2: MBP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2) | Phase 2: VCP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2) | Phase 2: VCP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2) | Phase 1: High Monetary Incentive (HMI) + VCP (Level 1 and Level 2) | Phase 1: High Monetary Incentive (HMI) + MBP (Level 1 and Level 2) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1 and Level 2) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1 and Level 2) | Phase 1: HMI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: HMI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2) | Phase 1: HMI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: HMI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2) | Phase 1: LMAI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: LMAI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2) | Phase 1: LMAI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: LMAI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2)
Number analyzed (Participants) | 105 | 93 | 114 | 144 | 126 | 117 | 14 | 11 | 12 | 17 | 10 | 11 | 11 | 13 | 12 | 13 | 13 | 16
units on a scale
  Baseline: number analyzed (Participants) | 105 | 93 | 114 | 144 | 126 | 117 | 14 | 11 | 12 | 17 | 9 | 9 | 11 | 12 | 11 | 13 | 13 | 15
  Baseline | 15.06 (4.67) | 15.30 (4.91) | 14.48 (5.33) | 15.14 (4.72) | 14.85 (4.79) | 15.09 (4.32) | 17.64 (3.77) | 20.91 (4.72) | 16.83 (4.93) | 16.59 (3.74) | 18.89 (3.48) | 16.67 (4.47) | 16.91 (3.65) | 16.67 (4.60) | 18.73 (4.86) | 15.23 (5.07) | 15.46 (5.27) | 16.80 (5.05)
  Week 6: number analyzed (Participants) | 94 | 82 | 105 | 130 | 108 | 106 | 11 | 10 | 8 | 15 | 9 | 9 | 10 | 12 | 8 | 9 | 11 | 11
  Week 6 | 5.55 (3.95) | 5.26 (3.97) | 10.57 (5.02) | 11.67 (5.03) | 11.15 (5.28) | 11.51 (5.09) | 7.18 (4.14) | 7.80 (3.85) | 7.00 (4.84) | 6.27 (4.40) | 12.56 (4.00) | 13.78 (5.78) | 11.30 (4.24) | 11.83 (5.64) | 14.00 (5.32) | 10.44 (6.25) | 11.00 (3.16) | 12.45 (5.50)
  Week 12: number analyzed (Participants) | 91 | 81 | 97 | 115 | 107 | 96 | 12 | 8 | 6 | 12 | 7 | 7 | 7 | 9 | 7 | 10 | 9 | 11
  Week 12 | 4.25 (4.15) | 3.88 (4.08) | 9.12 (6.05) | 9.91 (5.76) | 9.39 (5.98) | 10.43 (5.11) | 4.92 (3.92) | 7.38 (6.09) | 4.83 (1.94) | 5.42 (3.42) | 7.86 (3.34) | 9.57 (4.28) | 11.57 (5.32) | 11.33 (4.97) | 14.29 (4.82) | 11.30 (7.92) | 10.78 (5.65) | 9.64 (6.55)
Statistical Analysis 1: Comparison: Phase 2: Message-Based Psychotherapy (MBP; Level 1 and Level 2) vs Phase 2: Video-Chat Psychotherapy (VCP; Level 1 and Level 2); Mean difference comparing difference in average scores from baseline to week 6; Test type: Superiority; Mean Difference (Final Values) = 0.53
Statistical Analysis 2: Comparison: Phase 2: Message-Based Psychotherapy (MBP; Level 1 and Level 2) vs Phase 2: Video-Chat Psychotherapy (VCP; Level 1 and Level 2); Mean difference comparing difference in average scores from week 6 to week 12; Test type: Superiority; Mean Difference (Final Values) = 0.08
Statistical Analysis 3: Comparison: Phase 2: MBP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2) vs Phase 2: MBP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2); Mean difference comparing difference in average scores from baseline to week 6; Test type: Superiority; Mean Difference (Final Values) = 0.44
Statistical Analysis 4: Comparison: Phase 2: MBP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2) vs Phase 2: MBP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2); Mean difference comparing difference in average scores from week 6 to week 12; Test type: Superiority; Mean Difference (Final Values) = 0.31
Statistical Analysis 5: Comparison: Phase 2: VCP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2) vs Phase 2: VCP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2); Mean difference comparing difference in average scores from baseline to week 6; Test type: Superiority; Mean Difference (Final Values) = 0.12
Statistical Analysis 6: Comparison: Phase 2: VCP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2) vs Phase 2: VCP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2); Mean difference comparing difference in average scores from week 6 to week 12; Test type: Superiority; Mean Difference (Final Values) = 0.68

3. Secondary Outcome: Change in Generalized Anxiety Disorder (GAD-7)
Description: To assess for co-occurring anxiety, we will use the Generalized Anxiety Disorder-7 (GAD-7), a 7- item screener for generalized anxiety disorder (GAD). Participants rate on a scale of 0-3 how much they have experienced symptoms of GAD in the last two weeks. Total scores range from 0 to 21, with higher scores indicating greater severity of anxiety. The scale is a valid screener for GAD.
Time Frame: Change from Baseline GAD-7 at 6 weeks and 12 weeks after treatment starts
Population: All participants contributing data at baseline, week 6, or week 12. Overall number of participants analyzed includes total number of participants who contributed data at any relevant timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 2: Message-Based Psychotherapy (MBP; Level 1) | Phase 2: Video-Chat Psychotherapy (VCP; Level 1) | Phase 1: High Monetary Incentive (HMI) + VCP (Level 1) | Phase 1: High Monetary Incentive (HMI) + MBP (Level 1) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1)
Number analyzed (Participants) | 419 | 423 | 49 | 50 | 50 | 50
units on a scale
  Baseline: number analyzed (Participants) | 405 | 416 | 45 | 49 | 48 | 49
  Baseline | 12.22 (5.26) | 12.06 (5.04) | 14.76 (4.63) | 14.67 (5.12) | 13.27 (5.39) | 13.33 (5.08)
  Week 6: number analyzed (Participants) | 336 | 298 | 34 | 36 | 29 | 39
  Week 6 | 8.70 (5.12) | 8.21 (5.18) | 9.29 (4.51) | 10.11 (5.34) | 8.76 (5.67) | 8.77 (5.14)
  Week 12: number analyzed (Participants) | 293 | 281 | 30 | 30 | 24 | 33
  Week 12 | 6.98 (5.66) | 7.03 (5.55) | 7.17 (4.81) | 8.23 (5.70) | 9.04 (6.61) | 7.58 (5.70)

4. Other Pre Specified Outcome: Expectations About Treatment: Treatment Rationale Scale (TRS)
Description: Expectations about treatment can influence outcomes. To assess participant expectations, we will administer the Treatment Rationale Scale (TRS), a 4-item scale administered before the 2nd and last session. The scale assesses patient expectations about the success of treatment. Items are rated on a scale of 0 (not at all) to 10 (very). Total scores range from 0 to 40, with higher scores indicating better outcomes. 1) How logical does your Talkspace treatment seem to you? 2) How confident are you that the treatment will be successful in eliminating your depression? 3) How confident would you be in recommending the treatment to a friend with depression? 4) If you were extremely depressed, would you be willing to undergo such treatment?
Time Frame: Week 1
Population: Participants providing data on all items of the Treatment Rationale Scale at week 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 2: Message-Based Psychotherapy (MBP; Level 1) | Phase 2: Video-Chat Psychotherapy (VCP; Level 1) | Phase 1: High Monetary Incentive (HMI) + VCP (Level 1) | Phase 1: High Monetary Incentive (HMI) + MBP (Level 1) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1)
Number analyzed (Participants) | 383 | 348 | 41 | 41 | 37 | 43
units on a scale | 24.34 (9.38) | 26.98 (8.06) | 26.07 (7.75) | 25.71 (8.10) | 25.65 (7.88) | 24.74 (7.37)

5. Other Pre Specified Outcome: Experience of Care and Health Outcomes Survey (ECHO)
Description: The Experience of Care and Health Outcomes Survey (ECHO) items assess whether consumers received timely treatment, enough information to support self-management, and were involved in treatment as much as they wanted. ECHO is a reliable instrument with alpha = .85. For quality of care, participants rated an adapted version of item 28 of the Consumer Assessment of Healthcare Providers and Systems (CAHPS) ECHO survey: "In the past 4 weeks, using any number from 0 to 10, where 0 is the worst mental health care possible and 10 is the best mental health care possible, what number would you use to rate the mental health care you received from Talkspace?" Ratings range from 0 to 10. Higher scores indicate better quality of care received.
Time Frame: 10 weeks after treatment starts
Population: Participants randomized to a Level 2 condition contributing data at week 10.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Phase 2: MBP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2): Phase 2: This arm includes participants in MBP (Level 1) who did not respond to treatment by week 5. The Premium Plan (PP) intervention consists of MBP with monthly VCP (Level 2). The Premium Plan allows patients unlimited texting with their therapist and once a month, 30-45 minute video chat with the same therapist. This Level 2 intervention will serve as one of two augmentation "switch arms" for participants who do not respond to MBP or VCP alone by week 5.
- Phase 2: MBP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2): Phase 2: This arm includes participants in MBP (Level 1) who did not respond to treatment by week 5. The Ultimate Plan (UP) intervention consists of MBP with weekly VCP (Level 2). Like the Premium Plan, participants in the Ultimate Plan will have access to both unlimited MBP, but will be able to schedule weekly, 30-45 minute video chat with the same therapist. This Level 2 intervention will serve as one of two augmentation "switch arms" for participants who do not respond to MBP or VCP alone by week 5.
- Phase 2: VCP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2): Phase 2: This arm includes participants in VCP (Level 1) who did not respond to treatment by week 5. The Premium Plan (PP) intervention consists of MBP with monthly VCP (Level 2). The Premium Plan allows patients unlimited texting with their therapist and once a month, 30-45 minute video chat with the same therapist. This Level 2 intervention will serve as one of two augmentation "switch arms" for participants who do not respond to MBP or VCP alone by week 5.
- Phase 2: VCP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2): Phase 2: This arm includes participants in VCP (Level 1) who did not respond to treatment by week 5. The Ultimate Plan (UP) intervention consists of MBP with weekly VCP (Level 2). Like the Premium Plan, participants in the Ultimate Plan will have access to both unlimited MBP, but will be able to schedule weekly, 30-45 minute video chat with the same therapist. This Level 2 intervention will serve as one of two augmentation "switch arms" for participants who do not respond to MBP or VCP alone by week 5.
Arm/Group | Phase 2: Message-Based Psychotherapy (MBP; Level 1 and Level 2) | Phase 2: Video-Chat Psychotherapy (VCP; Level 1 and Level 2) | Phase 2: MBP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2) | Phase 2: MBP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2) | Phase 2: VCP (Level 1) to Premium Plan (MBP with monthly VCP; Level 2) | Phase 2: VCP (Level 1) to Ultimate Plan (MBP with weekly VCP; Level 2) | Phase 1: High Monetary Incentive (HMI) + VCP (Level 1 and Level 2) | Phase 1: High Monetary Incentive (HMI) + MBP (Level 1 and Level 2) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1 and Level 2) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1 and Level 2) | Phase 1: HMI + VCP (Level 1) to Augmentation Arm (MBP With Weekly VCP; Level 2) | Phase 1: HMI + VCP (Level 1) to Switch Arm (MBP With Monthly VCP; Level 2) | Phase 1: HMI + MBP (Level 1) to Augmentation Arm (MBP With Weekly VCP; Level 2) | Phase 1: HMI + MBP (Level 1) to Minimal Augmentation (MBP With Monthly VCP; Level 2) | Phase 1: LMAI + VCP (Level 1) to Augmentation Arm (MBP With Weekly VCP; Level 2) | Phase 1: LMAI + VCP (Level 1) to Switch Arm (MBP With Monthly VCP; Level 2) | Phase 1: LMAI + MBP (Level 1) to Augmentation Arm (MBP With Weekly VCP; Level 2) | Phase 1: LMAI + MBP (Level 1) to Minimal Augmentation (MBP With Monthly VCP; Level 2)
Number analyzed (Participants) | 92 | 80 | 98 | 118 | 105 | 98 | 9 | 10 | 7 | 11 | 9 | 8 | 9 | 9 | 7 | 7 | 8 | 9
units on a scale | 7.53 (1.97) | 8.09 (1.84) | 5.88 (2.57) | 6.11 (2.62) | 6.24 (2.47) | 6.42 (2.27) | 8.44 (1.59) | 5.90 (3.18) | 8.43 (1.13) | 5.64 (2.38) | 6.33 (2.65) | 6.63 (2.20) | 6.11 (2.15) | 4.67 (2.96) | 6.57 (1.72) | 8.29 (2.36) | 7.25 (2.66) | 6.22 (1.64)

6. Other Pre Specified Outcome: Working Alliance Inventory-Short Revised (WAI-SR)
Description: Participants rated therapeutic alliance using the Working Alliance Inventory-Short Revised (WAI-SR), a 12-item measure of therapeutic alliance (relationship between the consumer and therapist or coach) evaluating three domains: goals, tasks, and bond. Items are rated on a scale from 1 to 5. Total scores range from 12-60, with higher scores indicating a more effective therapeutic relationship. It is a reliable measure of alliance, with alpha = .92.
Time Frame: 10 weeks after treatment starts
Population: Participants randomized to a Level 2 condition contributing data at week 10.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 2: Message-Based Psychotherapy (MBP; Level 1 and Level 2) | Phase 2: Video-Chat Psychotherapy (VCP; Level 1 and Level 2) | Phase 2: MBP (Level 1) to Premium Plan (MBP With Monthly VCP; Level 2) | Phase 2: MBP (Level 1) to Ultimate Plan (MBP With Weekly VCP; Level 2) | Phase 2: VCP (Level 1) to Premium Plan (MBP With Monthly VCP; Level 2) | Phase 2: VCP (Level 1) to Ultimate Plan (MBP With Weekly VCP; Level 2) | Phase 1: High Monetary Incentive (HMI) + VCP (Level 1 and Level 2) | Phase 1: High Monetary Incentive (HMI) + MBP (Level 1 and Level 2) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1 and Level 2) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1 and Level 2) | Phase 1: HMI + VCP (Level 1) to Augmentation Arm (MBP With Weekly VCP; Level 2) | Phase 1: HMI + VCP (Level 1) to Switch Arm (MBP With Monthly VCP; Level 2) | Phase 1: HMI + MBP (Level 1) to Augmentation Arm (MBP With Weekly VCP; Level 2) | Phase 1: HMI + MBP (Level 1) to Minimal Augmentation (MBP With Monthly VCP; Level 2) | Phase 1: LMAI + VCP (Level 1) to Augmentation Arm (MBP With Weekly VCP; Level 2) | Phase 1: LMAI + VCP (Level 1) to Switch Arm (MBP With Monthly VCP; Level 2) | Phase 1: LMAI + MBP (Level 1) to Augmentation Arm (MBP With Weekly VCP; Level 2) | Phase 1: LMAI + MBP (Level 1) to Minimal Augmentation (MBP With Monthly VCP; Level 2)
Number analyzed (Participants) | 90 | 73 | 92 | 113 | 98 | 90 | 9 | 10 | 7 | 11 | 9 | 8 | 9 | 9 | 7 | 7 | 8 | 9
units on a scale | 47.70 (10.65) | 49.45 (9.73) | 38.28 (14.05) | 37.99 (14.38) | 41.78 (12.55) | 41.98 (10.92) | 50.56 (4.53) | 40.10 (17.97) | 49.29 (9.09) | 32.27 (9.90) | 35.78 (15.43) | 39.69 (12.16) | 34.11 (13.86) | 35.22 (12.42) | 37.86 (10.22) | 48.57 (12.65) | 43.00 (13.83) | 35.56 (8.38)

7. Other Pre Specified Outcome: Tailoring Variable - Response to Treatment
Description: To determine whether patients move to Level 2 treatment (starting at week 6), we will used clinician administered Patient Health Questionnaire-9 (PHQ-9) between weeks 3 to 5 of treatment. Response to treatment was defined as a PHQ-9 score less than 50% of the participant's baseline PHQ-9 score. Response to treatment was also evaluated via therapist feedback. Participants who responded to their Level 1 treatment assignment continued in that condition from weeks 6 to 12. Participants who did not respond to treatment were switched to either MBP with weekly VCP or to MBP with monthly VCP.
Time Frame: 6 weeks after treatment starts
Population: Includes participants assessed for Level 2 randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Message-Based Psychotherapy (MBP; Level 1) | Phase 2: Video-Chat Psychotherapy (VCP; Level 1) | Phase 1: High Monetary Incentive (HMI) + VCP (Level 1) | Phase 1: High Monetary Incentive (HMI) + MBP (Level 1) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1)
Number analyzed (Participants) | 363 | 336 | 37 | 37 | 37 | 46
Participants
  Responded to treatment | 105 | 93 | 15 | 11 | 12 | 17
  Did not respond to treatment | 258 | 243 | 22 | 26 | 25 | 29

8. Other Pre Specified Outcome: Treatment Use Variables: Number of Sessions Attended
Description: Phase 1: Number of distinct days of messaging plus number of live video sessions attended Phase 2: Number of sessions attended, defined as the number of sessions during which the client sent any messages or attended any video sessions, regardless of Level 1 condition (e.g., includes sessions during which participants in VCP only sent messages).
Time Frame: 12 weeks after treatment starts
Population: Includes participants who sent any number of messages or attended any number of video sessions.
Measure: Mean (Standard Deviation); unit: sessions
Groups:
- Phase 2: Message-Based Psychotherapy (MBP; Level 1): Phase 2 participants who respond to Message-Based Psychotherapy (MBP; Level 1) by 5 weeks of care will continue in this condition from weeks 6 to 12 (MBP; Level 2). Participants who do not respond to treatment by week 5 will be randomized to MBP+UP or MBP+PP (Level 2).
- Phase 2: Video-Chat Psychotherapy (VCP; Level 1): Phase 2 participants who respond to Video-Chat Psychotherapy (VCP; Level 1) by 5 weeks of care will continue in this condition from weeks 6 to 12 (VCP; Level 2). Participants who do not respond to treatment by week 5 will be randomized to VCP+UP or VCP+PP (Level 2).
Arm/Group | Phase 2: Message-Based Psychotherapy (MBP; Level 1) | Phase 2: Video-Chat Psychotherapy (VCP; Level 1) | Phase 1: High Monetary Incentive (HMI) + VCP (Level 1) | Phase 1: High Monetary Incentive (HMI) + MBP (Level 1) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1)
Number analyzed (Participants) | 377 | 358 | 51 | 51 | 50 | 50
sessions | 20.02 (16.30) | 16.10 (11.71) | 20.63 (13.00) | 70.33 (17.26) | 21.32 (80.27) | 22.54 (173.56)

9. Other Pre Specified Outcome: Treatment Use Variables: Number of Messages Sent
Description: Number of messages sent, regardless of condition (e.g., also includes number of messages sent by clients in VCP only).
Time Frame: 12 weeks after treatment starts
Population: Includes participants who sent any number of messages; excludes participants who sent no messages.
Measure: Mean (Standard Deviation); unit: number of messages
Arm/Group | Phase 2: Message-Based Psychotherapy (MBP; Level 1) | Phase 2: Video-Chat Psychotherapy (VCP; Level 1) | Phase 1: High Monetary Incentive (HMI) + VCP (Level 1) | Phase 1: High Monetary Incentive (HMI) + MBP (Level 1) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1)
Number analyzed (Participants) | 377 | 355 | 51 | 51 | 50 | 50
number of messages | 46.42 (55.63) | 26.19 (28.64) | 38.80 (38.45) | 70.33 (76.93) | 52.58 (80.27) | 109.04 (173.56)

10. Other Pre Specified Outcome: Treatment Use Variables: Time Between Patient and Psychotherapist Contact
Description: Time between patient and psychotherapist contact, defined as the number of days from client's Level 1 randomization date to the date of first psychotherapist message or video call. These data were available only for Phase 2.
Time Frame: 12 weeks after treatment starts
Population: Phase 2 participants who received a message from a psychotherapist or attended a video session.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Phase 2: Message-Based Psychotherapy (MBP; Level 1), MBP, MBP+UP, and MBP+PP (Level 2): Phase 2 participants who respond to Message-Based Psychotherapy (MBP; Level 1) by 5 weeks of care will continue in this condition from weeks 6 to 12 (MBP; Level 2). Participants who do not respond to treatment by week 5 will be randomized to MBP+UP or MBP+PP (Level 2).
- Phase 2: Video-Chat Psychotherapy (VCP; Level 1), VCP, VCP+UP, and VCP+PP (Level 2): Phase 2 participants who respond to Video-Chat Psychotherapy (VCP; Level 1) by 5 weeks of care will continue in this condition from weeks 6 to 12 (VCP; Level 2). Participants who do not respond to treatment by week 5 will be randomized to VCP+UP or VCP+PP (Level 2).
Arm/Group | Phase 2: Message-Based Psychotherapy (MBP; Level 1), MBP, MBP+UP, and MBP+PP (Level 2) | Phase 2: Video-Chat Psychotherapy (VCP; Level 1), VCP, VCP+UP, and VCP+PP (Level 2)
Number analyzed (Participants) | 420 | 425
days | 0.95 (3.16) | 0.93 (1.65)

ADVERSE EVENTS:
Time Frame: Phase 1: Adverse event data were collected through study completion, an average of 5 months. Phase 2: Adverse event data were collected through study completion, an average of 2 years.
Arm/Group | Phase 2: Message-Based Psychotherapy (MBP; Level 1 and Level 2) | Phase 2: Video-Chat Psychotherapy (VCP; Level 1 and Level 2) | Phase 2: MBP (Level 1) to Preimum Plan (MBP With Monthly VCP; Level 2) | Phase 2: MBP (Level 1) to Ultimate Plan (MBP With Weekly VCP; Level 2) | Phase 2: VCP (Level 1) to Preimum Plan (MBP With Monthly VCP; Level 2) | Phase 2: VCP (Level 1) to Ultimate Plan (MBP With Weekly VCP; Level 2) | Phase 1: High Monetary Incentive (HMI) + VCP (Level 1 and Level 2) | Phase 1: High Monetary Incentive (HMI) + MBP (Level 1 and Level 2) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1 and Level 2) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1 and Level 2) | Phase 1: HMI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: HMI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2) | Phase 1: HMI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: HMI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2) | Phase 1: LMAI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: LMAI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2) | Phase 1: LMAI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) | Phase 1: LMAI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2)
All-Cause Mortality (participants affected / at risk) | 0/485 | 0/484 | 0/114 | 0/144 | 0/126 | 0/117 | 0/55 | 0/54 | 0/52 | 0/54 | 0/10 | 0/12 | 0/13 | 0/13 | 0/12 | 0/13 | 0/13 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/485 | 1/484 | 0/114 | 0/144 | 0/126 | 0/117 | 0/55 | 1/54 | 0/52 | 0/54 | 0/10 | 0/12 | 0/13 | 0/13 | 0/12 | 0/13 | 0/13 | 0/16
Other Adverse Events (participants affected / at risk) | 0/485 | 0/484 | 0/114 | 0/144 | 0/126 | 0/117 | 0/55 | 0/54 | 0/52 | 0/54 | 0/10 | 0/12 | 0/13 | 0/13 | 0/12 | 0/13 | 0/13 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2: Message-Based Psychotherapy (MBP; Level 1 and Level 2) (N=485) | Phase 2: Video-Chat Psychotherapy (VCP; Level 1 and Level 2) (N=484) | Phase 2: MBP (Level 1) to Preimum Plan (MBP With Monthly VCP; Level 2) (N=114) | Phase 2: MBP (Level 1) to Ultimate Plan (MBP With Weekly VCP; Level 2) (N=144) | Phase 2: VCP (Level 1) to Preimum Plan (MBP With Monthly VCP; Level 2) (N=126) | Phase 2: VCP (Level 1) to Ultimate Plan (MBP With Weekly VCP; Level 2) (N=117) | Phase 1: High Monetary Incentive (HMI) + VCP (Level 1 and Level 2) (N=55) | Phase 1: High Monetary Incentive (HMI) + MBP (Level 1 and Level 2) (N=54) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + VCP (Level 1 and Level 2) (N=52) | Phase 1: Low Monetary and Alternative Incentive (LMAI) + MBP (Level 1 and Level 2) (N=54) | Phase 1: HMI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) (N=10) | Phase 1: HMI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2) (N=12) | Phase 1: HMI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) (N=13) | Phase 1: HMI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2) (N=13) | Phase 1: LMAI + VCP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) (N=12) | Phase 1: LMAI + VCP (Level 1) to Switch Arm (MBP with monthly VCP; Level 2) (N=13) | Phase 1: LMAI + MBP (Level 1) to Augmentation Arm (MBP with weekly VCP; Level 2) (N=13) | Phase 1: LMAI + MBP (Level 1) to Minimal Augmentation (MBP with monthly VCP; Level 2) (N=16)
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Participant self-admitted themselves for inpatient, psychiatric care (Phase 1: n=1, HMI+MBP [Level 1]; Phase 2: n=1, VCP [Level 1])

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT04513080/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT04513080/ICF_001.pdf